CLINICAL TRIAL: NCT05945264
Title: The Impact of a Culturally-based Live Music Intervention on the Metabolites and Metabolic Pathways Associated With Chronic Stress and the Risk of Pre-term Birth in Black Women
Brief Title: Music Intervention for Preterm Birth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Emory University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jacquelyn Taylor, Helen F. Pettit Professor of Nursing; Executive Director of Columbia Nursing's Center for Research of People of Color, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACYY0271; R01MD016899 (NIH); AAAU6262 (Other: Columbia University Irving Medical Center Institutional Review Board)
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Preterm Birth
Keywords: Chronic stress; Preterm birth; Black women stress; Metabolomics of chronic stress; Music and medicine; Music intervention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Intervention (MI) Group (Experimental): Music therapist will meet individually with each participant and provide music therapy content that reflects their culture and mood states.
  Interventions: Behavioral: Music Intervention (MI)
- Sham Control (SC) Group (Active Comparator): Music/Verbal therapist will meet individually with each participant but will provide verbal discourse only (i.e., no music therapy and verbal intervention only).
  Interventions: Other: Sham Control (SC)

INTERVENTIONS:
Behavioral: Music Intervention (MI) — The intervention will involve listening, playing and/or singing melodies or songs, that are meaningful to the participant, with interpretation/reflection on their relevance/capacity to alter stress.
  Arms: Music Intervention (MI) Group
Other: Sham Control (SC) — The intervention will be to support a woman to talk about anything she wants that is important to her.
  Other Names: Verbal intervention
  Arms: Sham Control (SC) Group

SUMMARY:
This study will test a music intervention (MI) versus a sham control (SC) arm which only includes a verbal intervention, to determine if the effects of the music intervention will reduce the biological impact of chronic stress among pregnant Black women, reduce preterm birth, and improve infant outcomes.

DETAILED DESCRIPTION:
Preterm birth occurs at unacceptably high rates in the United States, with Black women disproportionately affected. A long-recognized risk factor for preterm birth in this population is the relentless exposure to intersectional stress related to racial and sexual discrimination, poverty, and neighborhood disadvantage that Black women often experience from an early age. In this interdisciplinary study, the investigators bring together experts in preterm birth, music therapy, and metabolomics to address this health disparity by testing the efficacy of a live, culturally based music intervention to reduce the production of metabolites and metabolic pathways associated with chronic stress and thereby improve birth outcomes.

ELIGIBILITY:
Inclusion Criteria

* Aged 18 to 40 years
* Generally healthy pregnant women in the first trimester of pregnancy

Exclusion Criteria:

* Non-pregnant women
* Women with a chronic medical condition that could impact pregnancy health or duration
* Women regularly taking any medications other than prenatal vitamins

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-03-12 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-08-29 (Estimated)

PRIMARY OUTCOMES:
Score on the Perceived Stress Scale (PSS) | Week 1
  The Perceived Stress Scale (PSS) is a 10-item scale that was developed to measure the degree to which situations in one's life are appraised as stressful. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Scores range from 0 to 40 with higher scores indicating a worse outcome.
Score on the Perceived Stress Scale (PSS) | Week 5
  The Perceived Stress Scale (PSS) is a 10-item scale that was developed to measure the degree to which situations in one's life are appraised as stressful. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Scores range from 0 to 40 with higher scores indicating a worse outcome.
Score on the Perceived Stress Scale (PSS) | Week 10
  The Perceived Stress Scale (PSS) is a 10-item scale that was developed to measure the degree to which situations in one's life are appraised as stressful. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Scores range from 0 to 40 with higher scores indicating a worse outcome.
Mean Gestational Age | Up to 43 weeks
  Number of completed weeks/days of pregnancy will be collected and the mean will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Taylor, PhD, Principal Investigator — Columbia University; Joanne V. Loewy, DA, LCAT, MT-BC, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Louis Armstrong Center for Music and Medicine at Mount Sinai Health System, New York, New York
  - Columbia University Irving Medical Center/NewYork Presbyterian, New York, New York

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared, but de-identified composite data with be shared with authorized recipients at the end of the study.